CLINICAL TRIAL: NCT03484624
Title: Effect of Wearable Hip-Assist Robot on Reduction of Muscle Fatigue and Cardiopulmonary Metabolic Efficiency in Elderly Adults: A Preliminary Study
Brief Title: Effect of Wearable Hip-Assist Robot on Reduction of Cardiopulmonary Metabolic Efficiency in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-02-064
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2018-03

CONDITIONS: Gait
Keywords: Muscle; Fatigue; Wearable hip assist robot; Metabolic energy expenditure
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treadmill walking (Experimental): All subjects underwent measurements of muscle fatigue and respiratory metabolism energy during treadmill walking at a comfortable speed for 6 minutes and measured by three conditions (①NoGEMS-free gait, ②Torque off with GEMS, and ③Torque on with GEMS)
  Interventions: Device: Treadmill walking

INTERVENTIONS:
Device: Treadmill walking — All subjects underwent measurements of muscle fatigue and respiratory metabolism energy during treadmill walking at a comfortable speed for 6 minutes and measured by three conditions (①NoGEMS-free gait, ②Torque off with GEMS, and ③Torque on with GEMS)

SUMMARY:
The purpose of this study was to investigate the changes in muscle fatigue and respiratory metabolic energy expenditure during walking with wearable hip-assist robot (V3).

DETAILED DESCRIPTION:
The purpose of this study was to investigate the changes in muscle fatigue and respiratory metabolic energy expenditure during walking with wearable hip-assist robot (V3).

Metabolic energy expenditure and muscle fatigue are measured simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Elderly adults over age 65
* Those without a history of central nervous system disease

Exclusion Criteria:

* Those who have problems with walking due to problems such as visual field defects or fractures
* A person whose height is less than 140 cm or not more than 185 cm
* Body mass index BMI (body mass index) based on 35 or more obese
* Those with a cognitive problem that are difficult to understand and participate fully in this study
* Those who are at risk of falling when walking with serious dizziness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change on metabolic energy expenditure | 1 hour
  All subjects underwent measurements of respiratory metabolism energy during treadmill walking at a comfortable speed for 6 minutes and measured by three conditions (①NoGEMS-free gait, ②Torque off with GEMS, and ③Torque on with GEMS).
  Metabolic energy expenditure and muscle fatigue are measured simultaneously

SECONDARY OUTCOMES:
Change on muscle fatigue | 1 hour
  All subjects underwent measurements of muscle fatigue at a comfortable speed for 6 minutes and measured by three conditions (①NoGEMS-free gait, ②Torque off with GEMS, and ③Torque on with GEMS).
  Metabolic energy expenditure and muscle fatigue are measured simultaneously

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea